CLINICAL TRIAL: NCT00991315
Title: Assessment of Tumor Resistance and Stem Cells in Prostate Cancer
Brief Title: Collecting and Storing Blood and Tumor Tissue Samples From Patients Undergoing Prostatectomy or Transurethral Resection of the Prostate
Status: Terminated | Type: Observational
Why Stopped: Specimens are now collected through the BRS protocol.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Isaac Yi Kim, MD, PhD, MBA, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: 0220080275; P30CA072720 (NIH); 0220080275 (Other: IRB #); 080809 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be collected at time of TURP and will be deidentified and processed by standard procedures.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to collect material for study's to assess mechanisms of tumor progression, mechanisms of resistance, isolation of stem cells and biologic markers in tissue, serum and peripheral blood mononuclear cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing routine prostatectomy or transurethral resection of the prostate (TURP)

PATIENT CHARACTERISTICS:

5.1.1 Patient is undergoing routine prostatectomy or TURP.

5.1.2 Patient is ≥ 18 years old.

5.1.3 Patient must give informed consent.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing a routine prostatectomy or TURP (transurethral resection of the prostate) may be asked to participate
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2008-12-12 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Collection and freezing of tumor samples | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Kim, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States